CLINICAL TRIAL: NCT05222776
Title: Predictive Values for the Outcome of Ultrasound Guided Genicular Nerve Radiofrequency Ablation for Chronic Knee Pain
Brief Title: Predictive Values for the Outcome of Genicular Nerve Radiofrequency Ablation for Chronic Knee Pain
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Selin Guven Kose, Principal Investigator, Diskapi Teaching and Research Hospital
Other Study IDs: 122/03
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Researchers are trying to assess a predictive value or correlation between patient and procedural characteristics and outcome measures results after genicular nerve radiofrequency ablation.

DETAILED DESCRIPTION:
Genicular nerve radiofrequency stimulation procedure is an effective treatment for patients with chronic pain due to knee osteoarthritis; however, little is known about factors that predict procedure success. This study evaluated correlation between patient characteristics and procedural characteristics and pain improvement after ultrasound guided genicular nerve radiofrequency stimulation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient's 18 years or older
* Patients who recently underwent ultrasound guided genicular nerve radiofrequency (RF) procedure

Exclusion Criteria:

* lack of documentation of predictive factors to assess outcome
* Patients in whom adequate follow-up data was not available
* Patients who were prescribed a new analgesic drug or received concurrent treatments for different pain sources during the follow-up period, that could affect interpretation of genicular RF treatment results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent US guided radiofrequency procedures of the genicular nerves for chronic knee pain
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Pain assessed by NRS | Change from baseline pain score at 6 months
  A NRS involves asking the patient to rate his or her pain from 0 to 10 (11 point scale) with the understanding that 0 is equal to no pain and 10 is equal to worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: selin guven kose, MD, Principal Investigator — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)